CLINICAL TRIAL: NCT03563729
Title: Efficacy of Immunotherapy in Melanoma Patients With Brain Metastases Treated With Steroids
Brief Title: Melanoma Metastasized to the Brain and Steroids
Acronym: MEMBRAINS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM1807
Record Dates: First submitted 2018-06-06; First posted 2018-06-20 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Malignant Melanoma
Keywords: Immune therapy; checkpoint inhibitor; pembrolizumab; ipilimumab; nivolumab; steroid; brain metastasis; BRAF inhibitor; MEK inhibitor
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — pembrolizumab; Ipilimumab; Nivolumab; encorafenib; binimetinib; dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Six patients are enrolled in each arm. If clinical benefit is observed, each arm will be expanded to enroll a total of 20 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- B: Pembrolizumab (Prednisolone >10 mg) (Experimental): Intravenous infusion of pembrolizumab 2 mg/kg every third week for up to two years.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]
- C: Ipilimumab/nivolumab (Prednisolone 11-25 mg) (Experimental): Intravenous infusion of ipilimumab 3 mg/kg and nivolumab 1 mg/kg four times every three weeks in the induction phase and nivolumab 480 mg every four weeks in the maintenance phase for up to two years.
  Interventions: Drug: Ipilimumab Injection [Yervoy]; Drug: Nivolumab Injection [Opdivo]
- D: Ipilimumab/nivolumab (Prednisolone >25 mg) (Experimental): Intravenous infusion of ipilimumab 3 mg/kg and nivolumab 1 mg/kg four times every three weeks in the induction phase and nivolumab 480 mg every four weeks in the maintenance phase for up to two years.
  Interventions: Drug: Ipilimumab Injection [Yervoy]; Drug: Nivolumab Injection [Opdivo]
- E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg) (Experimental): Induction treatment with BRAF/MEK inhibitors (either the combination of encorafenib/binimetinib or dabrafenib/trametinib) orally for 28 days followed by intravenous infusion of ipilimumab 3 mg/kg and nivolumab 1 mg/kg four times every three weeks in the induction phase and nivolumab 480 mg every four weeks in the maintenance phase for up to two years.
  Interventions: Drug: Ipilimumab Injection [Yervoy]; Drug: Nivolumab Injection [Opdivo]; Drug: Encorafenib; Drug: Binimetinib; Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Alone
  Arms: B: Pembrolizumab (Prednisolone >10 mg)
Drug: Ipilimumab Injection [Yervoy] — In combination with nivolumab.
  Arms: C: Ipilimumab/nivolumab (Prednisolone 11-25 mg); D: Ipilimumab/nivolumab (Prednisolone >25 mg); E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)
Drug: Nivolumab Injection [Opdivo] — In combination with ipilimumab.
  Arms: C: Ipilimumab/nivolumab (Prednisolone 11-25 mg); D: Ipilimumab/nivolumab (Prednisolone >25 mg); E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)
Drug: Encorafenib — In combination with binimetinib
  Arms: E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)
Drug: Binimetinib — In combination with encorafenib
  Arms: E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)
Drug: Dabrafenib — In combination with dabrafenib
  Arms: E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)
Drug: Trametinib — In combination with trametinib
  Arms: E: BRAF/MEK -> ipi/nivo (prednisolone >10 mg)

SUMMARY:
This clinical trial is to clarify whether treatment with a checkpoint inhibitor alone (pembrolizumab) or two in combination (ipilimumab and nivolumab), results in clinical benefit for MM patients with brain metastases and in need of steroid treatment. Patients will be treated in four arms depending on steroid dose level at inclusion (> 10 < 25 mg prednisolone or > 25 mg prednisolone) and treatment (pembrolizumab alone or the combination of ipilimumab and nivolumab).

DETAILED DESCRIPTION:
Cancer immunotherapy with checkpoint inhibitors (CPI) has demonstrated significant response rates, with clinical responses of exceptional duration observed in pivotal clinical trials for multiple types of solid tumors. Results from clinical trials demonstrate a considerable survival benefit of CPI over standard treatments, leading to registration of CPI for lung-, head and neck-, bladder-, renal cancer, lymphomas and metastatic melanoma (MM). To date, CPI appear to hold the key for longterm survival - at least for patients treated in clinical trials.

Patients enrolled in pivotal clinical trials for immunotherapy of MM are highly selected and does not include patients with brain metastases. Small phase II studies lend support to CPI to yield responses in melanoma that has metastasized to the brain. However, a large proportion of patients that develop brain metastasis will require continued systemic treatment with steroids to alleviate symptoms from the central nervous system (CNS). This group of patients are not offered treatment with CPI, as it is generally assumed that steroid treatment hamper their clinical efficacy. Thus, this group of patients face a large unmet need.

Due to the immune inhibiting effects, steroids are used to manage immune-related adverse events (irAEs) induced by CPI treatment. However, patients receiving steroids in this context are still able to achieve and maintain clinical benefit even after stopping treatment.

It is not known whether steroid treatment at the time of initiation of CPI treatment diminishes the treatment effect, as patients in need of steroid treatment are generally excluded from clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic melanoma with radiologically verified brain metastasis
* Need for systemic steroid treatment (prednisolone > 10 mg daily; dexamethasone > 1.6 mg daily, hydrocortisone > 40 mg daily or equivalent) due to brain metastasis
* At least one measurable lesion according to RECIST version 1.1 guidelines
* Evaluable intracranial disease
* 18 years of age or older
* Performance status 0-2
* Able to undergo MRI with gadolinium contrast agent
* Adequate hematological and organ function
* No significant toxicity from previous cancer treatments (CTC<1)
* Women of childbearing potential: Negative serum pregnancy test and must use effective contraception. This applies from screening and until 6 months after treatment. Birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch are all considered effective contraceptives
* Men with female partner of childbearing potential must use effective contraception from screening and until 6 months after treatment. Effective contraceptives are as described above for the female partner. In addition documented vasectomy and sterility or double barrier contraception are considered effective contraceptives
* Signed statement of consent after receiving oral and written study information.
* Willingness to participate in the planned treatment and follow-up and capable of handling toxicities.
* For arm E specifically: Tumor cells must harbor BRAF mutation.

Exclusion Criteria:

* Another malignancy or concurrent malignancy unless disease-free for 3 years
* Ocular melanoma
* Neurological symptoms from brain metastases present at baseline despite steroid treatment, unless symptoms are related to prior surgery
* Known hypersensitivity to one of the active drugs or excipients
* Acute or chronic infections with HIV or hepatitis
* Any medical condition that will interfere with patient compliance or safety
* Prior treatment with anti-PD-1/PD-L1/PD-L2/CTLA-4 antibodies in the metastatic setting
* Prior systemic treatment with anti-PD-1/PD-L1/PD-L2/CTLA-4 antibodies in the adjuvant setting, unless completed more than 6 months before enrolment in this study
* Simultaneous treatment with other experimental drugs or other anti-cancer drugs
* Pregnant or breastfeeding females.
* For arm E specifically: Prior treatment with BRAF/MEK inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2028-06-06 (Estimated)

PRIMARY OUTCOMES:
6 months progression-free survival rate | 6 months
  Proportion of patients who did not progress or die within 6 months from commencing study treatment.
6 months overall survival rate | 6 months
  Proportion of patients who did not die within 6 months from commencing study treatment.

SECONDARY OUTCOMES:
Overall progression-free survival | 4 years
  Time from commencing study treatment to the date of progression or death.
Overall survival | 4 years
  Time from commencing study treatment to the date of death from any cause.
Overall response rate | 4 years
  Proportion of patients with an overall complete or partial response according to modified RECIST 1.1.
Extracranial response rate | 4 years
  Proportion of patients with an overall complete or partial response in extracranial lesions according to modified RECIST 1.1.
Intracranial response rate | 4 years
  Proportion of patients with an overall complete or partial response in intracranial lesions according to modified RECIST 1.1.
Intracranial clinical benefit rate | 4 years
  Proportion of patients with an overall complete, partial response or stable disease > 6 months according to modified RECIST 1.1.
Blood and tissue biomarkers of response and progression | 5 years
  Correlation of the baseline PD-L1 status, immune markers, genomics and other biomarkers in tumour tissue and blood with complete or partial response and at subsequent disease progressionanalyses of potential specific biomarkers predictive of response or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Troels H Borch, PhD, Principal Investigator — Center for Cancer Immune Therapy, Department of Hematology and Department of Oncology
Locations (3):
- Denmark (3):
  - Herlev Universityhospital, Herlev, Capital Region
  - Aarhus Universityhospital, Aarhus, Midt
  - Odense Universityhospital, Odense, Syd

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage of Center for Cancer Immune Therapy — https://www.herlevhospital.dk/ccit-denmark/Sider/default.aspx